CLINICAL TRIAL: NCT03824353
Title: Does Resilience to Childhood Adversity Improve With Social Intelligence Training
Brief Title: Social Intelligence Training in Midlife
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01AG048844 (NIH)
Record Dates: First submitted 2019-01-28; First posted 2019-01-31 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Social Skills; Social Interaction
MeSH Terms: conditions — Social Skills

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Intelligence Training (Experimental): The social intelligence training is delivered online to individuals in midlife (ages 40 and older). This is the sole active treatment condition within this RCT.
  Interventions: Behavioral: Social Intelligence Training
- Attention Control (Placebo Comparator): The attention control condition, known as The Healthy Living program provides information about different aspects of health.
  Interventions: Behavioral: The Healthy Living Program

INTERVENTIONS:
Behavioral: Social Intelligence Training — The social intelligence training consists of short 5-10 minute sessions organized into 7 modules designed to raise awareness of human nature and social relationships. The approach is based on evidence that social intelligence training is best advanced through interventions that modify key social cognitions regarding social engagement and enhance efficacy expectations regarding performance in social situations.
  Arms: Social Intelligence Training
Behavioral: The Healthy Living Program — A placebo condition delivered online which presents health-related information only.
  Arms: Attention Control

SUMMARY:
Childhood adversity leads to social difficulties, chronic illness, and early mortality for many, but not all adults: Some are resilient. The investigators will test whether an on-line program focused on enhancing social relationships for people in mid-life can increase the odds that those with a history of a troubled childhood will not suffer a greater loss in mental and physical health than those without those histories. The investigators findings will bring the field significantly closer to the day when low cost interventions can be offered that work to strengthen the capacities of people to overcome the challenges that arise from adverse treatment early in life.

DETAILED DESCRIPTION:
It is indisputable that health declines with age, and that the rate of decline is not the same for everyone. Many sources of accelerated risk of illness have been identified in prior research, and among the most reliable predictors of ill health are social stressors, including abusive social relations in childhood. Early life adversity may lead to poorer mental health and physical functioning in midlife through various pathways; among the most likely paths are social in origin, including troubled family relationships, heightened sensitivity to interpersonal stressors, and social isolation. Is it possible to interrupt this cause-effect pairing between early adversity and illness in later life? The investigators examine that question. Specifically, the investigators address whether the individual differences in risk attributable to childhood adversity are reversible through a social intelligence (SI) intervention for an established cohort of community residents who were part of a comprehensive study of biopsychosocial markers of resilience at Mid-Life. The investigators have three primary objectives in this research:

1. To examine whether an SI intervention can enhance the capacity for rewarding social relations, especially for individuals with a history of early life adversity.
2. To examine evidence for the investigator's hypothesis that intervention-related gains in the quality of social relationship will be responsible for the improvements in psychological, and physical functioning, and influence two bio-markers of health risk and resilience: interleukin 6 (IL-6) and DHEA-S.
3. To probe for individual differences in age, gender, history of abuse, personality, and genetic markers of risk that identify participants most responsive to the intervention.

To address these questions, an SI intervention will be delivered to a random-selected half of 220 middle-aged participants: Half with a history of child abuse and half who did not report abuse. The program is an on-line self-instructional series of videos with awareness exercises and behavioral practices designed to enhance fund of knowledge about relationships, increase skills, and enhance motivation to engage socially. In addition to charting social relations with daily diaries, the investigators will assess participants' social, psychological, and physical functioning at pre-test, post-test, three months, and six months following the intervention. The investigators hypothesize that the SI intervention will prompt lasting improvement in the ability to establish, maintain, and benefit from social relations in comparison to controls, which will lead to better psychological and physical functioning. The investigators will examine evidence for the hypothesis that the benefits of the intervention will be largest for individuals who have experienced greater early childhood adversity, as well as probe other individual differences in receptivity to the SI program that will inform future efforts to refine, test and disseminate this innovative program.

ELIGIBILITY:
Inclusion Criteria:

* Adult living in the US age 40 and older

Exclusion Criteria:

-

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change in social socio-emotion regulation. | Change will be assessed from baseline immeidately post intervention. This will be measured with four separate items that are on the same scale.
  Measured by standardized instruments in daily diary entries
Change in social intelligence | Change will be assessed from baseline immeidately post intervention, as well as at 3, and 6 month post intervention.
  Measured by a standardized instrument in the self-report questionnaires. We used the Tromso Social Intelligence Scale to assess social intelligence. The scale is comprised of 3 factors (social skills, social information processing, and social awareness). Each scale ranges from 1 to 5.
Change in social support and strain. | Change will be assessed from baseline immeidately post intervention, as well as at 3, and 6 month post intervention.
  Measured by a standardized instrument in the self-report questionnaires. We used the assessment tool described in Walen and Lachman (2000).
Change in well-being | Change will be assessed from baseline immeidately post intervention. A composite score will be created based on 16 items.
  Measured by standardized instruments in daily diaries

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Castro SA, Infurna FJ, Lemery-Chalfant K, Waldron VR, Zautra E. Are Daily Well-Being and Emotional Reactivity to Stressors Modifiable in Midlife?: Evidence from a Randomized Controlled Trial of an Online Social Intelligence Training Program. Prev Sci. 2023 Jul;24(5):841-851. doi: 10.1007/s11121-023-01492-7. Epub 2023 Mar 4. PMID 36870019
- [Derived] Castro SA, Infurna FJ, Lemery-Chalfant K, Waldron V, Zautra E. Can an online curriculum improve the daily socio-emotional lives of middle-aged adults exposed to childhood Trauma? Behav Res Ther. 2019 Jul;118:65-76. doi: 10.1016/j.brat.2019.03.012. Epub 2019 Mar 24. PMID 30999262